CLINICAL TRIAL: NCT05140148
Title: Promoting Recovery After STroke With Amantadine
Acronym: PRESTA
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Scott Kasner, MD, Professor of Neurology, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 849451
Record Dates: First submitted 2021-09-15; First posted 2021-12-01 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Stroke, Ischemic; Stroke Hemorrhagic
MeSH Terms: conditions — Ischemic Stroke; Hemorrhagic Stroke | interventions — Amantadine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator): placebo pill, twice daily
  Interventions: Drug: Placebo
- Amantadine (Active Comparator): 100 mg amantadine twice daily, or if 65 years or older once daily
  Interventions: Drug: Amantadine

INTERVENTIONS:
Drug: Amantadine — Amantadine is a antiviral drug and dopamine promoter that is currently approved by the FDA for the treatment of influenza A and Parkinson's Disease
  Arms: Amantadine
Drug: Placebo — placebo pills
  Arms: Placebo

SUMMARY:
The investigators aim to examine whether amantadine can help patients recover from stroke. This will be a blinded randomized clinical trial (RCT). Patients will be randomized post-ischemic or hemorrhagic stroke either to the placebo arm or amantadine arm. Patients will be on study drug or placebo for 1 month but will be enrolled for 3 months total. At various time points patients will be examined and fill out questionnaires to determine level of stroke recovery.

ELIGIBILITY:
Inclusion Criteria:

1. 18 to 85 years old, male and female
2. Modified Rankin Score (mRS)<=2 prior to stroke
3. Ischemic or hemorrhagic stroke as diagnosed by vascular neurologist or as proven on magnetic resonance imaging (MRI) or non-contrast head computed tomography NCHCT)
4. 24 hours to 3 weeks after stroke onset or time last known well prior to detection of symptoms
5. National Institute of Health Stroke Scale (NIHSS)>=3 and NIHSS<=15
6. Creatinine Clearance of greater than or equal to 60 mL/min using the Cockroft- Gault equation.
7. Have passed a swallow evaluation prior to drug administration
8. The patient is an acute rehabilitation candidate or candidate for the Homeward Stroke Program
9. Able to participate in administered tests

Exclusion Criteria:

1. Any degree of receptive aphasia
2. Moderate or severe expressive aphasia
3. Currently pregnant or plans to get pregnant
4. Currently breastfeeding
5. Any patient admitted with primary SubarachnoidH emorrhage (SAH )on either non-contrast head CT or MRI brain
6. Diagnosis of dementia or mild cognitive impairment prior to index stroke
7. Prior limb amputation
8. Currently prescribed or taking a primary anticholinergic medication
9. Currently enrolled in any other investigational pharmacologic or procedural clinical trial
10. Malignancy with active treatment
11. History of prior stroke with residual impairment
12. Current or prior neuroleptic use
13. History of suicidality or psychosis (The Columbia Suicide Severity Ratings Scale (C-SSRS) will be administered at the screening visit to assess depression and suicidal thoughts for subject eligibility. Any subjects who indicate severe depression or suicidal thoughts and/or attempts within the last year will not be eligible)
14. Prior history of seizures
15. Prior treatment with amantadine
16. Parkinson's disease
17. Amantadine allergy
18. Elevated liver function tests (aspartate aminotransferase and alanine aminotransferase above the upper limit of normal) -

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | Day 90
  Tolerability of the study drug will be assessed based on the proportion of patients who adherent with at least 80% of study medication.

SECONDARY OUTCOMES:
Global rating on the Stroke Impact Scale (SIS) | 90 days
  Patient reported measure of stroke recovery; Stroke Impact Scale has 59 items in 8 domains (each domain score ranges from 0-100) And a 9th domain that is an overall scale from 0-100. Each item in the first 8 domains is on a likert scale from 1-5 where 5 is better and 1 is worse
Total score on the National Institute of Health Stroke Scale (NIHSS) | 90 days
  Assessment for stroke deficits in patients; scores range from 0-42, with a higher score indicating more severe stroke symptoms
Digit Symbol Substitution Test (DSST) score | 90 Days
  Cognitive test; scores range from 0 to 100, with higher scores indicating higher cognitive function
Montreal Cognitive Assessment test (MOCA) score | 90 Days
  Cognitive test; scores range from 0 to 30, with higher scores indicating higher cognitive function
Patient Health Questionnaire (PHQ-9) score | 90 days
  Patient reported survey of depression symptoms; scores range from 0 to 27, with higher scores indicating higher levels of depression
Upper limb strength | 90 Days
  The upper limb strength for each subject with be measured using a hand dynamometer
Modified Rankin Score (mRS) | 90 days
  Assessment of post-stroke recovery; scores range from 0 to 6, with higher scores indicating more severe impairments on daily functioning

CONTACTS AND LOCATIONS:
Locations (1):
- The Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No